CLINICAL TRIAL: NCT02495506
Title: Transfusion Therapy in Patients Undergoing Cardiac Surgery in Combination With Late Withdrawal of Drug Induced Platelet Inhibition or Prolonged Extra-corporal Circulation Time
Brief Title: Transfusion of Cold-stored Platelet Concentrates
Acronym: 4CPLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/692
Record Dates: First submitted 2015-06-19; First posted 2015-07-13 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2018-09

CONDITIONS: Cardiovascular Disease Other; Bleeding; Surgery
Keywords: Cardiac surgery; bleeding; platelet transfusion
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cold stored platelets (Experimental): Intervention: Leukoreduced platelet concentrates stored at 4 degrees C for treatment of bleeding after Cardiac surgery
  Interventions: Other: Cold stored platelets
- Room temperature platelets (Active Comparator): Intervention: Leukoreduced platelet concentrates stored at 22 degrees C for treatment of bleeding after Cardiac surgery
  Interventions: Other: Room temperature platelets

INTERVENTIONS:
Other: Cold stored platelets — Intervention: Leukoreduced platelet concentrates stored at 4 degrees C for treatment of bleeding after Cardiac surgery. Storage time for RCT platelet concentrates are up to 7 days.
  Other Names: Trombocytes, Platelet concentrates
  Arms: Cold stored platelets
Other: Room temperature platelets — Intervention: Leukoreduced platelet concentrates stored at 22 degrees C for treatment of bleeding after Cardiac surgery. Storage time for RCT platelet concentrates are up to 7 days.
  Other Names: Trombocytes, Platelet concentrates
  Arms: Room temperature platelets

SUMMARY:
This study will investigate the effects of Leukocyte reduced cold-stored platelet transfusions used in treatment of immediate postoperative blood loss in patients undergoing thoracic surgery in combination with extracorporal circulation. Today platelet concentrates are stored at 22 degrees C .

This is a prospective, randomized, unblinded, non-inferiority two-arm study. Aim of study is to compare platelet function in bleeding patients transfused with leukoreduced platelet concentrates stored cold (4 degrees C) and in room temperature (22 degrees C). Storage time for RCT platelet concentrates are up to 7 days. Patients with expected time on extracorporal circulation more than 120 minutes and/or medical platelet inhibitors will be included.

Platelet function will be assessed by use of Multiplate Aggregometry, Thromboelastography (TEG) and/or Thromboelastometry (ROTEM). In addition post operative bleeding, and adverse events will be recorded.

After completion of recruitment of patients to RCT study of platelet stored cold for up to 7 days, a follow up prospective observational study of platelets stored cold for up to 14 days is performed.

Additonal information 2019, May 03: This trial was registered on Clinical Trials.gov with an original plan to use non-inferiority testing of between-group differences in platelet function. Due to lack of evidence needed to set acceptable tolerance margins for the non-inferiority testing, independent reviewers with expertise in clinical trial design recommended they be replaced by standard tests of superiority, commensurate with the early phase of the trial. Further, post-operative chest tube drainage was chosen as the primary outcome to better present the pilot study's focus on the control of clinically significant bleeding.

DETAILED DESCRIPTION:
This is a prospective, randomized, unblinded, non-inferiority two-arm study were Arm 1 patients will receive Leukocyte reduced cold-stored platelet concentrates and Arm 2 patients will receive leukoreduced room-temperature-stored (22 degrees C) platelet concentrates. Patients with expected time on extracorporal circulation more than 120 minutes and/or medical platelet inhibitors will be included.

The number of patients included is set to 20 patients in each arm, as there is not sufficient information available in the literature to conduct power calculations. The hypothesis is that cold stored platelets are not inferior to room temperature platelet concentrates.

Baseline patient data and information on intervention and post operative recovery will be collected from the Medical journals together with information on transfusion episodes and Blood Components. Blood samples will be retrieved from study participants at specific intervals: baseline, immediately after surgery, at arrival at ICU, before and after (every) platelet transfusion episode, 24 hours post operation, and if indicated, during hospital stay. Blood samples will be investigated for platelet function, coagulation parameters, hematologic parameters, and other risk factors for adverse events. If transfusion reactions occur, additional test of patient and the Blood Component(s) transfused will be performed. Samples will be collected and stored in the biobank for cytokines, complement and allergy analysis.

After completion of recruitment of patients to RCT study of platelet concentrates stored cold for up to 7 days, a follow up prospective observational study of platelets stored cold for up to 14 days is performed.

Additonal information 2019, May 03: This trial was registered on Clinical Trials.gov with an original plan to use non-inferiority testing of between-group differences in platelet function. Due to lack of evidence needed to set acceptable tolerance margins for the non-inferiority testing, independent reviewers with expertise in clinical trial design recommended they be replaced by standard tests of superiority, commensurate with the early phase of the trial. Further, post-operative chest tube drainage was chosen as the primary outcome to better present the pilot study's focus on the control of clinically significant bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing urgent/semiurgent thoracic surgery
* Expected long extracorporal time (>120 minutes) and/or use of dual platelet inhibition drugs
* Patients likely to require platelet transfusion
* Patients capable of providing informed consent

Exclusion Criteria:

* Patients who will not provide informed consent
* Patients with congenital coagulopathies or hemostatic disorders (von willebrands disease, hemophilia etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-03; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Chest drain output (postoperative bleeding) | 24 hours
  Information retrieved from Medical Journal

SECONDARY OUTCOMES:
Evidence of altered platelet function confirmed by Point-of-Care measurements | Up to 24 hours after surgery
  Evaluate in vitro changes in platelet function by use of the following Point-of-Care measurements; Multiplate whole blood impedance aggregometry, Thromboelastography, and ROTEM
Number of Blood Products transfused as a Measure of Bleeding | From date of inclusion during hospital stay, up to 4 weeks
  Information retrieved from Medical Journal
Number of Participants with thromboembolic events as a Measure of Safety | From date of procedure until the date of first documented event during hospital stay, up to 4 weeks
  Information retrieved from Medical Journal
Number of Participants with other adverse events as a Measure of Safety | From date of procedure until the date of first documented event during hospital stay, up to 4 weeks
  Information retrieved from Medical Journal
Number of Participants with transfusion complication as a Measure of Safety | From date of procedure until the date of first documented event during hospital stay, up to 4 weeks
  Information retrieved from Medical Journal
Hemoglobin value | From date of inclusion, daily during hospital stay, up to 4 weeks
  Information retrieved from Medical Journal
Hematocrit | Up to 24 hours after surgery
  Information retrieved from Medical Journal
Leukocyte count | Up to 24 hours after surgery
  Information retrieved from Medical Journal
Platelet count | From date of inclusion, daily during hospital stay, up to 4 weeks
  Information retrieved from Medical Journal
Fibrinogen | Up to 24 hours after surgery
  Information retrieved from Medical Journal
International normalized ratio (INR) | Up to 24 hours after surgery
  Information retrieved from Medical Journal
Activated Partial Thromboplastin time (APTT) | Baseline, up to 24 hours and at the date of first documented thromboembolic event during hospital stay, up to 4 weeks
  Information retrieved from Medical Journal
Allergy analysis as a Measure of Risk of transfusion complication | Baseline,and the date of first documented event during hospital stay, up to 4 weeks
  Information retrieved from Medical Journal
Complement analysis as a Measure of risk of transfusion complication | Baseline,and the date of first documented event during hospital stay, up to 4 weeks
  Information retrieved from Medical Journal

CONTACTS AND LOCATIONS:
Overall Officials: Geir Strandenes, MD, Principal Investigator — Haukeland University Hospital; Torunn Apelseth, MD/PhD, Study Director — Haukeland University Hospital; Einar Kristoffersen, MD/PhD, Study Chair — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No